CLINICAL TRIAL: NCT06152744
Title: Evaluation of Membrane Lung Function for Patients Receiving Venovenous Extracorporeal Membrane Oxygenation in High-altitude Regions
Brief Title: Evaluation of Membrane Lung Function in High-altitude Regions
Status: Recruiting | Type: Observational
Sponsor: Beijing Chao Yang Hospital (Other)
Collaborators: Affiliated Hospital of Qinghai University (Other)
Responsible Party: Principal Investigator, Rui Wang, Principal Investigator, Beijing Chao Yang Hospital
Other Study IDs: 2023-KE-1121
Record Dates: First submitted 2023-11-22; First posted 2023-12-01 (Actual); Last update posted 2025-06-17 (Actual); Status verified 2025-06

CONDITIONS: Extracorporeal Membrane Oxygenation; Membrane Lung Function; High Altitude
MeSH Terms: conditions — Altitude Sickness

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Biospecimen Retention: Samples With DNA — Arterial blood gas analysis, blood routine, liver and kidney function, coagulation, and BNP
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

GROUPS / COHORTS (2):
- High-altitude group
  Interventions: Other: Monitoring membrane lung function at different altitudes
- Low-altitude group
  Interventions: Other: Monitoring membrane lung function at different altitudes

INTERVENTIONS:
Other: Monitoring membrane lung function at different altitudes — The altitude in Beijing is 100m, while the altitude in Xining, Qinghai is 2600m. We will monitor the partial pressure of post-ML arterial oxygen in ECMO patients in these two locations and evaluate whether the normal values of membrane lung function are consistent in different altitudes.

SUMMARY:
Over the last 20 years, extracorporeal membrane oxygenation (ECMO) has been used to support adult patients with respiratory or cardiac failure who are unlikely to survive conventional treatment methods. ECMO circuit, pump, and oxygenator technology improvements permit safer perfusion for extended periods. The prolonged use of an ECMO circuit increases the risk of membrane lung (ML) dysfunction. The ML is responsible for taking in oxygen and removing carbon dioxide. The non-biologic surface of the ML triggers inflammatory and coagulation pathways, resulting in the formation of blood clots, breakdown of fibrin, and activation of white blood cells, which ultimately leads to ML dysfunction. Coagulation and fibrinolysis activation can cause systemic coagulopathy or hemolysis, and the deposition of blood clots can block blood flow. Moreover, the accumulation of moisture in the gas phase and the buildup of protein and cellular debris in the blood phase may contribute to shunt and dead-space physiology, respectively, impairing the exchange of gases. These three categories-hematologic abnormalities, mechanical obstruction, and inadequate gas exchange-account for most ML exchanges. Worsening oxygenation during ECMO should prompt quantification of oxygen transfer. ML exchange is indicated when the ML can no longer meet the patient's oxygen demand. The partial pressure of Post-ML arterial oxygen less than 200 mmHg is the most important consideration in this decision. In some high-altitude regions of China, ECMO treatment is also routinely conducted. The experiences above are derived from low-altitude areas, and whether they apply in high-altitude regions is still being determined. This study aimed to explore the significantly lower membrane lung oxygen uptake in high-altitude regions compared to low-altitude areas.

ELIGIBILITY:
Inclusion Criteria:

* Receiving ECMO support

Exclusion Criteria:

* Unable to obtain post-membrane blood gas
* Pregnancy
* Patients cannot receive anticoagulation
* Refusal to participate in the trial

Ages: 18 Years to 70 Years | Sex: All
Age Groups: Adult, Older Adult
Study Population: Patients who are supported by ECMO
Sampling Method: Non-Probability Sample
Enrollment: 40 (Estimated)
Dates: Start 2023-12-05 (Actual); Primary Completion 2025-12-30 (Estimated); Study Completion 2025-12-31 (Estimated)

PRIMARY OUTCOMES:
Initial assessment of membrane lung oxygen uptake | On the third day of ECMO support
  O2 content of post-ML blood - O2 content of pre-ML blood

SECONDARY OUTCOMES:
60-day mortality | After patients enrolled 60 days
  Mortality rate at 60 days of VV-ECMO support

CONTACTS AND LOCATIONS:
Overall Officials: Rui Wang, Dr., Study Director — Beijing Chao-Yang Hospital, Capital Medical University, Beijing, China
Locations (1):
- Beijing Chao-Yang Hospital, Beijing, Beijing Municipality, China

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Zakhary B, Vercaemst L, Mason P, Antonini MV, Lorusso R, Brodie D. How I approach membrane lung dysfunction in patients receiving ECMO. Crit Care. 2020 Nov 30;24(1):671. doi: 10.1186/s13054-020-03388-2. No abstract available. PMID 33256824